CLINICAL TRIAL: NCT03649984
Title: Implementation of the Symptom Navi© Program for Cancer Patients in Ambulatory Services: A Cluster-randomized Pilot Study (Symptom Navi© Pilot Study)
Brief Title: Implementation of the Symptom Navi© Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuela Eicher (Other)
Responsible Party: Sponsor-Investigator, Manuela Eicher, Prof. Dr., University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Symptom Navi© Pilot Study
Record Dates: First submitted 2018-05-30; First posted 2018-08-28 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Cancer
Keywords: Symptom-management; Outpatients; Nurse-led intervention; Implementation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: cluster-randomized waitlist design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptom Navi© Program (Experimental): Nurses provide two semi-structured consultation to facilitate basic symptom self-management of patients based in the Symptom Navi© Flyers
  Interventions: Behavioral: Symptom Navi© Program
- Standard care (No Intervention): Standard care including information about treatment, potential side effects and expected symptoms under treatment with or without additional written material following the established procedure at the centre.

INTERVENTIONS:
Behavioral: Symptom Navi© Program — Trained nurses provide two semi-structured patient education consultations with Symptom Navi© Flyers. Patients will use the Symptom Navi© Flyers individually at home.
  Arms: Symptom Navi© Program

SUMMARY:
The Symptom Navi© Program is a program to support symptom self-management of 16 core symptoms frequently experienced by patients in outpatient oncology units.The current study aims to pilot test the implementation of the Symptom Navi© Program under real-life conditions by evaluating procedures, testing preliminary effectiveness and assessing potential unintended effects using a cluster-randomised waitlist design complemented by qualitative methods.

DETAILED DESCRIPTION:
Patients treated in cancer outpatient settings in Switzerland have high unmet care needs, especially in the domain of self-management of symptoms. The Symptom Navi© Program was developed to support symptom self-management of 16 core symptoms frequently experienced by patients in outpatient oncology units. The acceptability and feasibility of the Symptom Navi© Program was supported by a qualitative study with 10 cancer patients who received semi-structured patient consultations and subsequently used the Symptom Navi© Flyers at home.

The overall objective of the current study is to pilot test the implementation of the Symptom Navi© Program under real-life conditions. The aims are to evaluate procedures, to test preliminary effectiveness and to assess potential unintended effects using a cluster-randomised waitlist design complemented by qualitative methods. The unit of randomization are the participating cancer outpatient centres with each centre representing a cluster. Intervention cluster will provide the Symptom Navi© Program, control clusters will provide usual care for symptom-management.

ELIGIBILITY:
Inclusion Criteria for patients:

* age ≥ 18 years
* newly diagnosed with cancer within 15 weeks prior to informed consent signature
* planned to receive first cycle of their first-line pharmacological anti-cancer treatment in an outpatient centre (intravenous, oral or subcutaneous)
* signed informed consent

Exclusion Criteria for patients:

* not sufficiently literate in German language to understand written information or follow an interview
* recurrence of cancer disease
* cared by a palliative care team
* being treated solely with surgical or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported symptom interference with daily function | Change from baseline to 16 weeks
  Symptom interference with daily function in the affective and activity subdimension scores of the MD Anderson Symptom Inventory (MDASI)

SECONDARY OUTCOMES:
Reach of intervention in terms of proportion of eligible vs. participating patients | Up to 16 weeks
Change in patient-reported self-efficacy | Change from baseline to 16 weeks
  Self-efficacy assessed by the Self-Efficacy for Managing Chronic Disease (SES6G)
Change in patient-reported symptom severity | Change from baseline to 16 weeks
  Symptom severity assesssed by the MD Anderson Symptom Inventory (MDASI)
Change in patient-reported quality of nursing care | Change from baseline to 16 weeks
  Quality of nursing care assessed by the Patient-Reported Chemotherapy Indicators of Symptoms and Experiences (PR-CISE)
Incidence of Intervention-Emergent Adverse Events | Up to 16 weeks
  Adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Eicher, Prof. Dr., Study Director — UniLausanne
Locations (9):
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Gynäkologisches Tumorzentrum Universitätsspital Basel, Basel
  - Oncocare, Klinik Engeried Bern, Bern
  - Kantonsspital Graubünden, Chur
  - Hôpital fribourgeois - Meyriez-Murten / Tagers, Murten/Morat
  - Tumor- und Brustzentrum ZeTuP Rapperswil, Rapperswil
  - Rundum Onkologie am Bahnhofpark Sargans, Sargans
  - Solothurner Spitäler AG - Kantonsspital Olten / Bürgerspital Solothurn, Solothurn
  - Spital STS AG - Thun, Thun

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bana M, Ribi K, Peters S, Kropf-Staub S, Naf E, Zurcher-Florin S, Stoffel B, Blaeuer C, Borner M, Malin D, Biber R, Betticher D, Kuhn-Bachler T, Cantoni N, Seeger T, Butikofer L, Eicher M; Symptom Navi Program Group. Pilot Testing of a Nurse-Led Basic Symptom Self-management Support for Patients Receiving First-Line Systemic Outpatient Anticancer Treatment: A Cluster-Randomized Study (Symptom Navi Pilot Study). Cancer Nurs. 2021 Nov-Dec 01;44(6):E687-E702. doi: 10.1097/NCC.0000000000000995. PMID 34507338
- [Derived] Bana M, Ribi K, Kropf-Staub S, Naf E, Schramm MS, Zurcher-Florin S, Peters S, Eicher M. Development and implementation strategies of a nurse-led symptom self-management program in outpatient cancer centres: The Symptom Navi(c) Programme. Eur J Oncol Nurs. 2020 Feb;44:101714. doi: 10.1016/j.ejon.2019.101714. Epub 2019 Dec 20. PMID 31954227
- [Derived] Bana M, Ribi K, Kropf-Staub S, Zurcher-Florin S, Naf E, Manser T, Butikofer L, Rintelen F, Peters S, Eicher M. Implementation of the Symptom Navi (c) Programme for cancer patients in the Swiss outpatient setting: a study protocol for a cluster randomised pilot study (Symptom Navi(c) Pilot Study). BMJ Open. 2019 Jul 9;9(7):e027942. doi: 10.1136/bmjopen-2018-027942. PMID 31289075